CLINICAL TRIAL: NCT02696642
Title: An Open Label Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of Anetumab Ravtansine in Subjects With Mesothelin-expressing Advanced Solid Cancers and Different Stages of Concurrent Hepatic or Renal Impairment
Brief Title: Phase I Study of Anetumab Ravtansine in Hepatic or Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18327; 2015-003897-33 (EudraCT Number)
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Neoplasms
Keywords: mesothelin-expressing advanced solid cancers
MeSH Terms: conditions — Neoplasms | interventions — anetumab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Experimental): Anetumab ravtansine was given at 6.5 mg/kg body weight (BW) as a 1 hour intravenous (IV) infusion once every 3 weeks (Q3W) for subjects with adequate hepatic and renal function.
  Interventions: Drug: Anetumab ravtansine (BAY94-9343)
- mild HI group (Experimental): Anetumab ravtansine was given at 6.5 mg/kg BW as a 1 hour IV infusion Q3W for subjects with mild hepatic impairment (HI).
  Interventions: Drug: Anetumab ravtansine (BAY94-9343)
- moderate HI group (Experimental): Anetumab ravtansine was given at 6.5 mg/kg BW as a 1 hour IV infusion Q3W for subjects with moderate hepatic impairment (HI).
  Interventions: Drug: Anetumab ravtansine (BAY94-9343)
- moderate RI group (Experimental): Anetumab ravtansine was given at 6.5 mg/kg BW as a 1 hour IV infusion Q3W for subjects with moderate renal impairment (RI).
  Interventions: Drug: Anetumab ravtansine (BAY94-9343)

INTERVENTIONS:
Drug: Anetumab ravtansine (BAY94-9343) — All subjects received anetumab ravtansine 6.5 mg/kg BW (body weight) once every three weeks

SUMMARY:
To characterize the safety, tolerability, pharmacokinetics and immunogenicity of anetumab ravtansine in subjects with advanced solid cancers and with different degrees of hepatic or renal impairment

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years
* Histologically or cytologically confirmed, locally advanced or metastatic solid cancers known to express mesothelin on the tumor cell surface (e.g. predominantly epithelial [>=50% tumor component] pleural or peritoneal mesothelioma, epithelial ovarian cancer [including the fallopian tube or primary peritoneal], adenocarcinoma of the pancreas, triple-negative adenocarcinoma of the breast, non-small-cell adenocarcinoma of the lung, endometrial cancer, serous uterine cancer, gastric cancer [including the gastro-esophageal junction], colon cancer, cholangiocarcinoma, thymic carcinoma, etc.). Subjects with resected primary cancers who have documented metastases or local recurrence are eligible.
* Subjects must have no standard therapy available, or have actively refused standard therapy
* Subjects must meet the criteria for one of the 4 treatment groups:

  * Group A: Adequate hepatic and renal function (controls)
  * Group B: Mild hepatic impairment, i.e. Grade A according to the Child-Pugh Classification (total score of 5 or 6) and adequate renal function
  * Group C: Moderate hepatic impairment, i.e. Grade B according to the Child-Pugh Classification (total score of 7, 8 or 9) and adequate renal function
  * Group D: Moderate renal impairment, i.e. eGFR (estimated glomerular filtration rate) <60 and ≥30 mL/min per 1.73 m*2 and hepatic function better than, or equal to mild impairment according to the Child-Pugh Classification (total score ≤6)
* Adequate bone marrow function
* Life expectancy of at least 12 weeks
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1 (control and mild hepatic impairment groups), or 0-2 (moderate hepatic impairment and moderate renal impairment groups)

Exclusion Criteria:

* Subjects who have a previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study, except cervical carcinoma in situ, treated basal cell carcinoma, superficial noninvasive bladder tumors or any previous cancer curatively treated >3 years before the start of anetumab ravtansine
* Subjects who have new or progressive brain or meningeal or spinal metastases
* Subjects who have Gilbert's syndrome or other benign congenital hyperbilirubinemia are not eligible for the mild or moderate hepatic impairment or moderate renal impairment groups.
* Subjects who have a history or current evidence of bleeding disorder, i.e. any hemorrhage/bleeding event of CTCAE (Common Terminology Criteria for Adverse Events) Grade ≥2 bleeding within 4 weeks before the start of anetumab ravtansine
* Subjects who have a history or current evidence of uncontrolled cardiovascular disease or hypertension.
* Fridericia-corrected QT interval (QTcF) >480 ms, heart rate ≥100 beats per minute (bpm) or ≤45 bpm, LVEF (left ventricular ejection fraction) <50%
* Subjects with corneal epitheliopathy or any eye disorder that may predispose the subjects to drug-induced corneal epitheliopathy or may interfere with diagnosis of treatment-emergent corneal epitheliopathy at the investigator's discretion in consultation with an ophthalmologist.
* Subjects who have received systemic anticancer therapy (except pemetrexed, cisplatin, carboplatin and topical or intracavitary treatments with negligible absorption in systemic circulation ) within 4 weeks before the start of anetumab ravtansine, or within 5 half-lives of the anticancer agent before the start of anetumab ravtansine, whichever is longer. Mitomycin C or nitrosoureas must be excluded within 6 weeks before the start of anetumab ravtansine.
* Subjects who have received radiotherapy within 4 weeks before the start of anetumab ravtansine
* Use of drugs that, in the opinion of the investigator, have a strong potential for renal or hepatic toxicity within 2 weeks before the start of anetumab ravtansine until the EoT visit.
* Use of strong cytochrome P450 3A4 (CYP3A4) inhibitors or strong CYP3A4 inducers within 2 weeks before the start of anetumab ravtansine until the EoT visit
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) and significant abnormalities in safety assessments related to anetumab ravtansine (BAY94-9343) in each of the 4 treatment groups | After the first application of the study drug up until the safety follow up visit, i.e., 30-35 days after the last dose of the study drug.
AUC for antibody drug conjugate (ADC), total antibody (TA), derivative 4 of maytansine (DM4), and S methyl derivate of DM4 (DM4-Me) after single (first) dose administration of anetumab ravtansine (BAY94-9343) in Cycle 1 | From pre-dose until 504 hours post dose during cycle 1
AUC(0-tlast) for ADC, TA, DM4 and DM4-Me after single (first) dose administration of anetumab ravtansine (BAY94-9343) in Cycle 1 | From pre-dose until 504 hours post dose during cycle 1
Cmax for ADC, TA, DM4 and DM4-Me after single (first) dose administration of anetumab ravtansine (BAY94-9343) in Cycle 1 | From pre-dose until 504 hours post dose during cycle 1

SECONDARY OUTCOMES:
Cmax,md for ADC, TA, DM4 and DM4-Me in Cycle 3 | From pre-dose until 504 hours post dose during cycle 3
AUC(0-tlast)md for ADC, TA, DM4 and DM4-Me in Cycle 3 | From pre-dose until 504 hours post dose during cycle 3
Number of subjects with positive immunogenicity results for anti anetumab ravtansine (BAY94-9343) antibodies (anti drug antibody [ADA]) | From pre-dose on Day1 of Cycle 1 until the safety follow-up visit, i.e., 30-35 days after the last dose of the study drug
Number of subjects with positive immunogenicity results for anetumab ravtansine (BAY94-9343) neutralizing antibody (NAB) | From pre-dose on Day1 of Cycle 1 until the safety follow-up visit, i.e., 30-35 days after the last dose of the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- France (7):
  - Caen
  - Dijon
  - Lille
  - Lyon
  - Marseille
  - Saint-Herblain
  - Toulouse
- Chisinau, Moldova

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/